CLINICAL TRIAL: NCT02890004
Title: A Prospective, Observational Registry of Patient With Subarachnoid Hemorrhage in Neurocritical Care Unit
Brief Title: Observational Study of Patients With Subarachnoid Hemorrhage
Acronym: ProReSHA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0561
Record Dates: First submitted 2016-08-24; First posted 2016-09-07 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: Subarachnoid Hemorrhage; Neurointensive care; Observational registry
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, observational study aim to identify :

* Prognostic factor of patients with subarachnoid haemorrhage in neuro intensive care unit
* The impact of standard therapeutic used (surgery, embolization ; medical treatment of vasospasm ; treatment of complications like hyponatremia, stress myocardiopathy, …)

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the unit of investigator with subarachnoid hemorrhage, whatever the etiology, is included in their prospective registry
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2020-03-16 (Estimated); Study Completion 2020-03-16 (Estimated)

PRIMARY OUTCOMES:
Survival | at day 0
Survival | at 6 months
Survival | at 12 months

SECONDARY OUTCOMES:
Neurological outcome with the Glasgow Coma Scale (GCS) score | at day 0
Neurological outcome with the Glasgow Coma Scale (GCS) score | at 6 months
Neurological outcome with the Glasgow Coma Scale (GCS) score | at 12 months
Neuropsychological outcome with the Montreal Cognitive Assessment (MoCA) score | at day 0
Neuropsychological outcome with the Montreal Cognitive Assessment (MoCA) score | at 6 months
Neuropsychological outcome with the Montreal Cognitive Assessment (MoCA) score | at 12 months
Brain lesions with MRI | at day 0
Brain lesions with MRI | at 6 months
Brain lesions with MRI | at 12 months
delay of apparition of hyponatremia | on alternte days after Day 0
  Natremia in standard blood sample, Natremia is routinelly evaluated on alternte days, and more if required.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DAILLER, MD, Principal Investigator — Service de réanimation neurologique Hospices Civils de Lyon
Locations (1):
- Service de réanimation polyvalente neurologique Hôpital Neurologique HCL, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chardon N, Nourredine M, Ledochowski S, Kurland NT, Dailler F, Ritzenthaler T, Nougier C, Balanca B. Trajectory of mean platelet volume changes after aneurysmal subarachnoid hemorrhage in patients with or without delayed cerebral ischemia. Sci Rep. 2024 Oct 24;14(1):25122. doi: 10.1038/s41598-024-75587-8. PMID 39448701